# Macrophage Markers in Periodontal and Peri-implant Health and Disease (NCT05242354)

### Study protocol

## Background

CD80, CD163 and CD206 have been used in prior research in specifying macrophage phenotypes in periodontal and peri-implant tissues (1-5). However, there are no previously published studies on total gingival levels of CD163, CD206 and CD80 comparing peri-implantitis, periodontitis, peri-implant health and periodontal health.

### Primary objective

• to reveal the differences in CD163, CD206 and CD80 tissue levels between peri-implantitis, periodontitis, peri-implant health and periodontal health

# Subject population (n=36)

- applied to Biruni University between March-December 2021
- systemic healthy and ≥18 years-old non-smokers with no regular medicine intake who are willing to
  participate
- no antibiotics or anti-inflammatories for the last 3 months
- not pregnant, not in lactation
- according to the healthy or diseased groups:
  - diagnosed with peri-implantitis or generalized Stage III periodontitis at least one BoP+ periodontal/peri-implant pocket with a PPD of 6 10 mm
  - periodontally healthy in need of crown lengthening, gingivectomy, tooth extraction or dental implant application (having no pockets with PPD ≥ 4 mm and having a full mouth score of BoP < 10%)
  - having a submerged implant, which is partially exposed and has no visible signs of inflammation

### Clinical data

Probable pocket depth, indirect clinical attachment loss, and bleeding on probing from six sites of all teeth / implants

### Tissue samples

- Periodontitis and peri-implantitis samples during non-surgical therapy with a single stroke using Gracey curette
- Healthy peri-implant mucosa during implant exposure surgery with an incisional biopsy
- Healthy gingiva during the corresponding treatment with a crestal incision reaching the bottom of the crevice.

### Quantification of CD163, CD206 and CD80

- grinding of tissues with a high-speed tissue homogenizer
- protein determination with a commercial protein determination kit
- immunoblot analysis of each sample according to their total protein counts
- quantification of the band intensities

### Statistics

- Kruskal-Wallis test to reveal the differences of CD163, CD206 and CD80 levels (arbitrary units) between groups (peri-implantitis, periodontitis, peri-implant health, periodontal health)
- Mann Whitney U test pairwise comparison of groups showing significant differences according to Kruskal-Wallis test.
- Chi-square qualitative variables
- p < 0.05 significant

#### References

1. Galarraga-Vinueza ME, Obreja K, Ramanauskaite A, et al (2021) Macrophage polarization in peri-implantitis lesions. Clin Oral Invest 25:2335–2344.

- 2. Fretwurst T, Garaicoa-Pazmino C, Nelson K, et al (2020) Characterization of macrophages infiltrating periimplantitis lesions. Clin Oral Impl Res 31:274–281.
- 3. Thorbert-Mros S, Larsson L, Berglundh T (2015) Cellular composition of long-standing gingivitis and periodontitis lesions. J Periodont Res 50:535–543.
- 4. Fretwurst T, Müller J, Larsson L, et al (2021) Immunohistological composition of peri-implantitis affected tissue around ceramic implants—A pilot study. J Periodontol 92:571–579.
- Almubarak A, Tanagala KKK, Papapanou PN, et al (2020) Disruption of Monocyte and Macrophage Homeostasis in Periodontitis. Front Immunol 11:330.